CLINICAL TRIAL: NCT04445376
Title: Effect of Aerobic Exercises on Cardio-respiratory Fitness and Quality of Life in Recovered COVID 19 Recovered Patients.
Brief Title: Effect of Physical Therapy Exercises on Cardiorespiratory Fitness Level in COVID19 Patients After Recovery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Physiotherapist, Government College University Faisalabad
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 313
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Cardiorespiratory fitness
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Ventilatory) (Experimental): Breathing Exercise and Aerobic Training will be provided to all the patients.The training session will be given 3 days a week.
  Interventions: Other: Physical Exercises
- Intervention (Non ventilatory) (Experimental): Breathing Exercise and Aerobic Training will be provided to all the patients.The training session will be given 3 days a week.
  Interventions: Other: Physical Exercises

INTERVENTIONS:
Other: Physical Exercises — Aerobic Training and Breathing Exercises.

SUMMARY:
In some patients, lung function declined by about 20 to 30% after recovery. Computer tomography of COVID-19 patients revealed a ground glass opacity in both lungs. We will measure the Cardiorespiratory fitness according to American College of Sports medicine guidline and provide physiotherapy exercise to the patients to measure the improvement.

DETAILED DESCRIPTION:
In December 2019, the first reports emerged of a novel severe acute respiratory syndrome (SARS) coronavirus 2 (SARS-CoV-2) in Wuhan, China. The virus, which causes atypical pneumonia progressing to acute lung injury and acute respiratory distress syndrome (ARDS) in some individuals, was named COVID-19. The burden of fibrotic lung disease following SARS-CoV-2 infection is likely to be high; therefore, given the scale of the pandemic, the global burden of fibrotic lung disease will probably increase considerably. The aim of this study is to check the cardiorespiratory fitness level and the effect of Physical therapy intervention to improve the Cardiorespiratory fitness level in patients recovered from COVID-19. Quality of life has also been affected due to COVID19 due to decreased Cardiorespiratory fitness level, and this study also aims to improve the quality of life of people recovered from COVID19.

ELIGIBILITY:
Inclusion Criteria:

* Recovered from COVID 19 disease (PCR report).
* Sub-normal performance as compared to normative data.
* Do not have any Respiratory Problem.
* Consent to participate in the study.
* Able to understand and perform the exercise.
* Age from 18 to 75.
* Dyspnea due to COVID19.
* Modified Borg Dyspnea Scale score at least 2 but less than 7.

Exclusion Criteria:

* Not suffered from COVID 19.
* Respiratory Problem.
* Resting Blood Pressure greater than 160/100 instead of taking medicine
* Greater than 1-month post COVID19 Recovery.
* Cardiorespiratory comorbidities which limit participation in exercise.
* Any Musculoskeletal problem which limit participation in Training.
* Other cardiovascular morbidity which would limit exercise tolerance (heart failure, abnormal blood pressure responses or ST-segment depression > 2mm, symptomatic aortic stenosis, complex arrhythmias).
* Unstable angina
* Orthostatic blood pressure decrease of >20 mmHg with symptoms
* Hypertropic cardiomyopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 5 weeks
  To measure the cardio-respiratory fitness.
Modified Borg Dyspnea Scale | 5 weeks
  It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal.

SECONDARY OUTCOMES:
SF-36 QUESTIONNAIRE | 5 weeks
  The SF-36 questionnaire consists of 36 items, which are used to calculate eight subscales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The first four scores can be summed to create the physical composite score (PCS), while the last four can be summed to create the mental composite score (MCS). Scores for the SF-36 scales range between 0 and 100, with higher scores indicating a better HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Ishtiaq Ahmed, DPT, Principal Investigator — Government College University
Locations (1):
- Bin Inam Rehabilitation Center., Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George PM, Wells AU, Jenkins RG. Pulmonary fibrosis and COVID-19: the potential role for antifibrotic therapy. Lancet Respir Med. 2020 Aug;8(8):807-815. doi: 10.1016/S2213-2600(20)30225-3. Epub 2020 May 15. PMID 32422178
- [Background] Belli S, Balbi B, Prince I, Cattaneo D, Masocco F, Zaccaria S, Bertalli L, Cattini F, Lomazzo A, Dal Negro F, Giardini M, Franssen FME, Janssen DJA, Spruit MA. Low physical functioning and impaired performance of activities of daily life in COVID-19 patients who survived hospitalisation. Eur Respir J. 2020 Oct 15;56(4):2002096. doi: 10.1183/13993003.02096-2020. Print 2020 Oct. PMID 32764112